CLINICAL TRIAL: NCT04208568
Title: Gallbladder Counting on Epigastric Site;A Randomized Trial Comparing Postoperative Pain After Gallbladder Retrieval From Umblical and Epigastric Port Site in Laproscopic Cholecystectomy
Brief Title: Comparison of Postoperative Pain After Gallbladder Retrieval From Umbilical and Epigastric Ports.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baqai Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: Muhammad Danish Muneeb
Record Dates: First submitted 2019-12-16; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Cholelithiasis
MeSH Terms: conditions — Cholelithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gallbladder retrieval from umbilical port (Active Comparator): Gallbladder retrieved from 10 mm umbilical port.
  Interventions: Procedure: Laparoscopic cholecystectomy
- Gallbladder retrieval from epigastric port (Active Comparator): Gallbladder retrieved from 10 mm epigastric port.
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Four ports laparoscopic cholecystectomy under general anaesthesia

SUMMARY:
To know the association of postoperative pain after gallbladder removal from umbilical port site versus epigastric portsite, after four ports laparoscopic cholecystectomy,and the epigastric port site was found to be friendly for the patients in terms of less pain after gallbladder removal from this site after surgery.

DETAILED DESCRIPTION:
Objective: To know the association of postoperative pain after gallbladder removal from umbilical port site versus epigastric port site, after four ports laparoscopic cholecystectomy.

Randomized controlled trial was performed during 1-year period from January 2017 till January 2018, at a private hospital setup. Both male and female patients, with age group 18 and above, in years, were considered, who were planned four ports laparoscopic cholecystectomy after typical cholelithiasis. Those patients with polyps , mucocele or empyema in gallbladder or perforated gallbladder requiring emergency surgery were omitted from the study. The patients were randomly selected, 65 in which gallbladder was removed from umbilical region (group A) and 65 from epigastric region (group B) respectively. Determination of postoperative pain was done on day one, at the time of release from the hospital and at follow-up time one-month post-surgery, with the help of Numerical Analogue Scale (NAS).

ELIGIBILITY:
Inclusion Criteria:

* All healthy patients without cholecystitis

Exclusion Criteria:

* Acute cholecystits, mucocoele, empyema, carcinoma, peritonitis, ASA 3 and 4

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
comparison of postoperative pain after laparoscopic cholecystectomy between umbilical and epigastric port sites, using Numerical Analogue Scale (NAS). | 1 year
  Numerical Analogue Scale (NAS) was used to measure the pain score.

IPD SHARING:
Plan to Share IPD: No